CLINICAL TRIAL: NCT01263730
Title: Tai Chi Training for Treating Depressed Chinese Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Albert Yeung, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2008P000262
Record Dates: First submitted 2010-12-06; First posted 2010-12-21 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tai Chi Training (Active Comparator): The active group will be given 12 weeks of tai chi training
  Interventions: Behavioral: Tai Chi
- Waitlist control group (No Intervention): There is a waitlist control group that will receive the training following a 12 week no treatment period of time

INTERVENTIONS:
Behavioral: Tai Chi — Tai Chi training consists of a sequence of slow, soft, and graceful movements derived from the martial arts. It is considered as a moving form of yoga and meditation combined. Tai Chi has been considered as one form of oriental healing arts, like acupuncture, which fosters the circulation of this 'chi' or energy within the body.
  Arms: Tai Chi Training

SUMMARY:
The goal of this research is to evaluate whether Tai Chi merits further investigation as a non-pharmacological therapy in the treatment of Major Depressive Disorder (MDD). Specifically, this waitlist-controlled study will gather preliminary data evaluating the effectiveness of Tai Chi training as treatment for patients with MDD or a history of MDD, including patients who continue to be depressed despite taking antidepressants and patients who choose not to take antidepressants due to fear of side effects and/or for personal reasons. To test this hypothesis the investigators will compare physical and psychological parameters of a control group and an intervention group, at baseline (Week 0), at the midpoint (Week 6), and at the end of 12 weeks of Tai Chi training.

DETAILED DESCRIPTION:
When a first line treatment for depression fails, clinicians often choose to increase the dosage, or augment with a second agent, prior to considering switching agents altogether (Rosenbaum et al, 1995). Combination of an SSRI/SNRI with other agents such as tricyclic antidepressants (TCAs) or lithium are examples of popular strategies (Fava et al, 1994). In many instances, augmentation with multiple psychotropic agents may not be desirable, because of risk of side effects or drug-drug interactions.

In view of their benign adverse effect profiles, non-pharmacological interventions such as psychotherapy and mind-body intervention have been used to augment treatment for treatment resistant depressed patients. Preliminary studies have shown that meditation is beneficial for the treatment of depression (Smith et al., 2007; Sephton et al., 2007; Finucane and Mercer, 2006; Astin et al., 2003; Speca et al., 2000).

Tai Chi training consists of a sequence of slow, soft, and graceful movements derived from the martial arts. It is considered as a moving form of yoga and meditation combined. Tai Chi has been considered as one form of oriental healing arts, like acupuncture, which fosters the circulation of this 'chi' or energy within the body. By doing so, the health and vitality of the person are enhanced. Tai Chi, with its slow movement synchronized to the person's breathing, has been known to lead to a calm and tranquil mind when the person is focused on the precise execution of these exercises.

ELIGIBILITY:
General Inclusion criteria

* Men and women between the ages of 18 and 65 years;
* Satisfy DSM-IV criteria for current Major Depressive Disorder (MDD), or have a history of MDD, prior to the initiation of Tai Chi treatment, as determined by the SCID interview;
* Have not had Tai Chi treatment training and have not started other forms of mind/body intervention in the past 3 months.

General Exclusion criteria

* Patients with primary diagnosis other than MDD and/or do not have a history of MDD;
* Conditions that may make it difficult to conclusively determine that depressive symptoms are the result of MDD or having a history of MDD and not some other condition, including any form of substance abuse or dependence within the last 6 months, relevant medical conditions that may be the medical basis of a depression including epilepsy, history of an abnormal EEG, severe head trauma, or stroke;
* Medical conditions that would preclude entry into a clinical trial, including serious uncontrolled medical conditions (e.g. poorly controlled diabetes, severe congestive heart failure), or other medical conditions that have not been stable for a minimum of 3 months);
* Confounding treatments, such as current ongoing treatment other than what is provided by South Cove for depression; plans to receive confounding treatments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Depressive Symptoms | 12 weeks of Tai Chi Training
  We will be looking for a decrease in depressive symptoms at the mid- (week 6) and post- (week 12) time point following Tai Chi training as compared to the baseline (week 0).

SECONDARY OUTCOMES:
Psychological questionnaires, specifically the Quality of Life Enjoyment questionnaire. | 12 weeks of Tai Chi Training
  We will compare psychometric questionnaire results pre-(wk 0), mid- (wk 6), and post- (wk 12) Tai Chi training. The questionnaires administered include the Hamilton Depression Rating Scale, Clinical Global Inventory, Patient Health Questionnaire, Beck Depression Inventory, Quality of Life Enjoyment and Satisfaction, Expectations Tai Chi training on depression, International Physical Activity, and Mimet's Multidimensional Scale of Perceived Social Support.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Yeung, MD, Principal Investigator — Massachusetts General Hospital; John W. Denninger, MD, Study Director — Massachusetts General Hospital; Herbert Benson, MD, Study Director — Massachusetts General Hospital; Gregory Fricchione, MD, Study Director — Massachusetts General Hospital
Locations (1):
- South Cove, Boston, Massachusetts, United States